CLINICAL TRIAL: NCT04020848
Title: Observe Alternating Hemiplegia of Childhood (OBSERV-AHC) Prospective Observational Natural History and Therapy Study
Brief Title: Observe Alternating Hemiplegia of Childhood (OBSERV-AHC) Study
Acronym: OBSERV-AHC
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0199; 2019-A00860-57 (Other: ID-RCB)
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Alternating Hemiplegia
MeSH Terms: conditions — Alternating hemiplegia of childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Alternating Hemiplegia of Childhood (AHC): Patients who fit the Aicardi Alternating Hemiplegia of Childhood clinical criteria of any age. The Aicardi Criteria are six (Heinzen et al 2015). (1) Paroxysmal hemiplegia episodes. (2) Bilateral hemiplegia or quadriplegia episodes. (3) Other paroxysmal manifestations, such as abnormal eye movements, nystagmus, strabismus, ataxia, dystonia, choreoathetosis, tonic spells, or autonomic disturbances. (4) Evidence of permanent neurological dysfunction, which can manifest as cognitive impairment, developmental delay, and/or persistent motor deficits such as spastic diplegia/quadriplegia, hypotonia, ataxia, choreoathetosis, or dystonia. (5) Sleep relieves symptoms, although attacks may resume soon after awakening. (6) First signs of dysfunction occur prior to the age of 18 months.
  Patients having some but not all the above criteria and have the mutation in ATP1A3 gene can be included.
  Interventions: Other: Review of past medical history, clinical exam, and electroencephalogram, polysomnography and urine samples of melatonin and pupillometry.; Other: The patients' parents have to complete the VINELAND II adaptive behavior scales scoring, The Sleep Disturbance Scale for Children (SDSC) and Horne & Ostberg Circadian Typology Questionnaire

INTERVENTIONS:
Other: Review of past medical history, clinical exam, and electroencephalogram, polysomnography and urine samples of melatonin and pupillometry. — Review of past medical history; review of paroxysmal events; identification of presence of seizures & epilepsy & epilepsy classification; characterization of the non-paroxysmal features; degree of paroxysmal, non-paroxysmal disability indices; Vineland II adaptive behavior scales scoring; behavioral evaluation; presence of a genetic mutation; pharmacological treatments already used; AHC paroxysmal events assessement during the time of study; patient calendar for the follow up of events, for the follow up of epileptic seizures; whether, or not, there was occurrence of a serious or potentially life-threatening event (status epilepticus, apnea requiring intervention, or death) during time of study; growth and somatic complaints; further information concerning family history & comorbidities; past instrumental & biochemical investigations (ECG, cardiac ultrasound results if done as part of patient's follow-up); electroencephalogram; polysomnography; urine samples of melatonin ; pupillometry
Other: The patients' parents have to complete the VINELAND II adaptive behavior scales scoring, The Sleep Disturbance Scale for Children (SDSC) and Horne & Ostberg Circadian Typology Questionnaire — Sleep Disturbance Scale for Children ; Horne & Ostberg Circadian Typology Questionnaire

SUMMARY:
Alternating Hemiplegia of Childhood (AHC) is a rare and serious disease that is in need of effective, and hopefully even curative, therapies. Afflicted patients suffer from severe paralyzing crises, often excruciatingly painful muscle spasms, severe often life threatening epileptic seizures, and frequently severe developmental and psychiatric/psychological disabilities. Based on the repeated input from family organizations and from professionals, as expressed at the London 2016 ATP1A3 in Disease meeting, there are urgent clinical research needs for AHC that are essential to better understand the disease, evaluate its treatment options and plan for future controlled clinical trials.

The goal of the study is to evaluate different parameters involved in the evolution of the AHC. The investigating team's hypothesis is that the evolution is variable so it aims to evaluate the factors which could contribute to the progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

- Patients who fit the Aicardi Alternating Hemiplegia of Childhood clinical criteria of any age. The Aicardi Criteria are six :

* Paroxysmal hemiplegia episodes.
* Bilateral hemiplegia or quadriplegia episodes.
* Other paroxysmal manifestations, such as abnormal eye movements, nystagmus, strabismus, ataxia, dystonia, choreoathetosis, tonic spells, or autonomic disturbances.
* Evidence of permanent neurological dysfunction, which can manifest as cognitive impairment, developmental delay, and/or persistent motor deficits such as spastic diplegia/quadriplegia, hypotonia, ataxia, choreoathetosis, or dystonia.
* Sleep relieves symptoms, although attacks may resume soon after awakening.
* First signs of dysfunction occur prior to the age of 18 months.

Exclusion Criteria:

* Patients who do not have a mutation of the ATP1A3 gene and having only some of the above criteria
* Patients and / or their parents / legal guardian having provided their opposition to the study.
* Incapacity of patient / parent or other referent adult to participate in the prospective phase of observation of different paroxysmal events of the disease and in the scoring of the Vineland II adaptive behavior scales.
* Diagnosis of another disease, which could explain the presence of symptoms mentioned in the criteria of Aicardi.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alternating Hemiplegia of Childhood (AHC)
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
final index compared to the initial index of non-paroxysmal disability | 1 year: Inclusion Visit up to 1 year visit
  The aim is to study the modification of the final index compared to the initial index of non-paroxysmal disability in order to evaluate the parameters that influence its evolution.
  The non-paroxysmal disability index is calculated from different variables : ability to walk independently, presence of a behavioral disorder, presence and degree of communication disorders, abnormality of global motor skills, abnormality of fine motor skills, movements disorders, intellectual deficiency. The study also aims to evaluate the sleep architecture in AHC

CONTACTS AND LOCATIONS:
Overall Officials: Eleni PANAGIOTAKAKI, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon Department of Clinical Epileptology, Sleep Disorders and Functional Neurology in Children, Bron, France